CLINICAL TRIAL: NCT00192660
Title: Analysis of Lipodystrophy in HIV-Infected Individuals A Prospective, Non-randomised, 48 Week Study of the Effect of PI Containing and Non-PI Containing Antiretroviral Regimens on the Expression of Adipocyte Specific Genes, Protein Levels and Cellular Structure in HIV-infected Individuals, Naive to Therapy, Who Are Starting Therapy for the First Time
Brief Title: HIV Infection And Metabolic Abnormalities Protocol 1 (HAMA001)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kirby Institute (Other Government)
Collaborators: St Vincent's Hospital, Sydney (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HAMA 001 Version 6; R01HL065953-01 (NIH)
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2012-04-12 (Estimated); Status verified 2012-04

CONDITIONS: HIV-Associated Lipodystrophy Syndrome; Cardiovascular Disease
Keywords: HIV; Metabolic abnormality; Lipodystrophy; Cardiovascular disease; Treatment Naive; Treatment Experienced; HIV Infections
MeSH Terms: conditions — HIV-Associated Lipodystrophy Syndrome; Cardiovascular Diseases; Lipodystrophy; HIV Infections | interventions — Lamivudine; Stavudine; Didanosine; Zidovudine; Tenofovir; abacavir; efavirenz; Nevirapine; Indinavir; Saquinavir; amprenavir; Ritonavir; Nelfinavir; tipranavir; Enfuvirtide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Lamivudine
Drug: Stavudine
Drug: Didanosine
Drug: Zidovudine
Drug: Tenofovir
Drug: Abacavir
Drug: Efavirenz (EFV)
Drug: Nevirapine
Drug: Indinavir
Drug: Saquinavir
Drug: Amprenavir
Drug: Ritonavir
Drug: Nelfinavir
Drug: Tipranavir
Drug: enfuvirtide (T20)

SUMMARY:
This is a prospective, non-randomised, 48 week study of the effect of protease inhibitor (PI) containing and non-PI containing antiretroviral regimens on the expression of adipocyte specific genes, protein levels and cellular structure in HIV-infected individuals, naive to therapy, who are starting therapy for the first time.

DETAILED DESCRIPTION:
Antiretroviral medications, used to treat HIV infection, cause side effects. These include changes in composition of fat throughout the body (loss in some areas and accumulation in others), elevations in blood lipids and abnormalities in glucose metabolism. The resulting syndrome is known as "HIV associated lipodystrophy" or HIVLD. In HIV negative populations, such abnormalities in lipid and glucose metabolism are associated with an increased risk of developing cardiovascular disease (CVD). The aim of this study is to characterize the changes that occur in body composition and metabolism with antiretroviral treatment and compare them to changes in fat tissue structure and function and surrogate markers for cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* Age >18.
* Be able to provide written consent to perform in the trial.
* HIV antibody positive at time of entry to the study.

Specific to HIV Infection and Metabolic Abnormalities Protocol 1 (HAMA) part A only:

* Be naive to antiretroviral medication.

Specific to HAMA part B only:

* Have had a minimum total exposure to antiretroviral medications (to include drugs from more than one drug class) of 48 weeks at time of recruitment.
* Have had a minimum of 48 weeks interval since completion of HAMA part A.

Exclusion Criteria:

* Any history of, or ongoing, mental or physical condition (including suspected or known diagnosis of ischaemic heart disease), which, in the opinion of the investigator, would impede the subject's ability to participate in the trial.
* Prior use of growth hormone or glucocorticoid or anabolic steroid products within the previous six months.
* Prior use of supraphysiological doses of testosterone or oestrogen replacement therapy within the previous year.
* Alcohol or substance abuse which in the opinion of the investigator would affect the patients ability to participate in the trial.
* Prior use of any retinoid-containing compound within the previous six months.
* Abnormal coagulation.
* Previous allergic reaction or known allergy to local anaesthetic.
* Previous or concomitant use of medications, which, in the opinion of the investigator, would affect the subject's ability to participate in all activities involved in the trial.
* Any grade-three laboratory abnormality recorded from screening bloods, which, in the opinion of the investigator, would impede the subject's ability to safely complete all study requirements.
* Any finding on screening clinical examination, which, in the opinion of the investigator, would impede the subject's ability to participate in the rest of the trial.
* Pregnancy

Specific to HAMA part A only:

* Prior use of anti-retroviral agents (including protease inhibitors, nucleoside or non-nucleoside reverse transcriptase inhibitors, investigational antiretroviral agents or fusion inhibitors). Entry of individuals who have had previous antiretroviral therapy as part of post exposure prophylaxis will be at the discretion of the study investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2003-02; Primary Completion 2006-10 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
To investigate changes in adipocyte structure and function in HIV-infected individuals treated with antiretroviral therapy

SECONDARY OUTCOMES:
To correlate changes in adipocyte function with changes in body composition and metabolic parameters in individuals beginning their first antiretroviral regimen
To examine changes in adipocyte function in HIV-infected volunteers both prior to and after initiation of treatment in order to determine changes arising directly as a result of therapy
To investigate changes in adipocyte function in pre-treated HIV-infected volunteers with and without established signs of HIVLD in order to determine if changes in function correlate with particular phenotypes such as lipoatrophy or buffalo hump

CONTACTS AND LOCATIONS:
Overall Officials: Andrew D Carr, MD, Principal Investigator — St. Vincents Hospital Sydney Limited; David A Cooper, MD, Study Director — The National Centre in HIV Epidemiology and Clinical Research, Sydney
Locations (1):
- St. Vincent's Hospital, Sydney, New South Wales, Australia

REFERENCES:
- See also: National Centre in HIV Epidemiology and Clinical Research Homepage — http://www.med.unsw.edu.au/nchecr/